CLINICAL TRIAL: NCT07333014
Title: Adapted Visual Safety Plan for Autistic Youth (VSP-AY) to Address Self-harm, Suicidal Ideation, and Suicide Behaviors: : A Pilot Randomized Controlled Trial
Brief Title: Adapted Visual Safety Plan for Autistic Youth (VSP-AY) to Address Self-harm, Suicidal Ideation, and Suicide Behaviors
Acronym: VSP-AY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Management Academic Studies (Other)
Collaborators: Geha Mental Health Center (Other); University of Haifa (Other); Tel Aviv University (Other); Reichman University (Other); University of Nottingham (Other); La Trobe University (Other); Deakin University (Other); Bournemouth University (Other)
Responsible Party: Principal Investigator, Ella Sarel-Mahlev, PhD. Senior Lecturer Rank, College of Management Academic Studies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VSP-AY-2025-Pilot
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; Suicidal Ideation; Suicidal Behavior; Self-Injurious Behavior; Depression
Keywords: Autistic adolescents; Visual safety plan; Self-harm; NSSI; Mental health intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Suicidal Ideation; Self-Injurious Behavior; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An Interventional study VSP-AY (Experimental): Participants receive the Visual Safety Plan for Autistic Youth (VSP-AY) intervention in addition to treatment as usual. VSP-AY is an autism-adapted safety planning tool incorporating linguistic modifications (concrete language, explicit examples), visual supports (color-coding, progressive revelation), and developmental appropriateness for adolescents.
  Interventions: Behavioral: Adapted Visual Safety Plan for Autistic Youth (VSP-AY) to Address Self-harm, Suicidal Ideation, and Suicide Behaviors
- No Intervention: Treatment as Usual (No Intervention): Participants receive standard mental health care at Geha Mental Health Center without the VSP-AY intervention.

INTERVENTIONS:
Behavioral: Adapted Visual Safety Plan for Autistic Youth (VSP-AY) to Address Self-harm, Suicidal Ideation, and Suicide Behaviors — The Visual Safety Plan for Autistic Youth (VSP-AY) is an autism-adapted suicide prevention tool delivered as a visual card-based system with supporting materials. The intervention includes two main sections: intrapersonal strategies (recognizing warning signs, internal coping skills) and interpersonal strategies (social contacts, professional resources, means safety).
  VSP-AY uses visual cards with color-coding to guide the safety planning process. Participants choose where to begin, accommodating individual preferences and processing styles. Each component offers multiple phrasing options and includes concrete examples drawn from autistic individuals with lived experience, making content accessible and relevant.
  Supporting materials include: writing sheets where participants document their personalized strategies; communication cards for different settings (home, school, community) with explicit guidance on what to do and what not to do during suicidal crisis moments; visual supports
  Arms: An Interventional study VSP-AY

SUMMARY:
This pilot randomized controlled trial will recruit 90 autistic adolescents aged 13-18 years with recent suicidal thoughts or behaviors from Geha Mental Health Center in Israel. Participants will be randomly assigned in a 1:1 ratio to either (1) the intervention group receiving the Visual Safety Plan for Autistic Youth (VSP-AY) plus standard care, or (2) the control group receiving treatment as usual without VSP-AY. Mental health professionals delivering VSP-AY will complete a 6-hour training with ongoing supervision throughout the study. Outcomes will be assessed at three timepoints: baseline (T0), immediately post-intervention (T1), and one-month follow-up (T2). The study will evaluate feasibility through recruitment and completion rates, acceptability through satisfaction questionnaires and qualitative interviews, and preliminary effectiveness through standardized measures of suicidal ideation (Columbia Suicide Severity Rating Scale), non-suicidal self-injury (NSSI-AT), and depression (Children's Depression Inventory).

DETAILED DESCRIPTION:
Background Autistic individuals face a significantly higher risk of suicide compared to the general population, with recent meta-analyses consistently showing rates up to three times higher across various groups, including general autistic samples and those without any intellectual disability. Other meta-analytical data indicate pooled prevalence rates of lifetime suicidal ideation at 37.2% and suicide attempts at 15.3% among autistic individuals.

This increased risk is mainly due to co-occurring psychiatric conditions. Autistic individuals with any psychiatric disorder have 3.55 times higher odds of self-harm compared to those without such conditions. These psychiatric conditions are consistently linked to poorer health outcomes, reduced quality of life, and increased suicidal behaviors.

While suicide among autistic adults has received substantial research attention, autistic youth have been less studied. However, emerging evidence shows that this higher risk also applies to younger groups. Epidemiological research indicates that autistic youth aged 10-19 years have 4.27 times higher rates of suicide deaths and 2.83 times higher rates of suicide attempts compared to their non-autistic peers. A Korean study of school-aged children also found increased rates of parent-reported suicidal ideation among those with autism spectrum disorder compared to neurotypical peers. Similarly, a UK cohort study showed that youth with social communication challenges had significantly higher risks for self-harm with suicidal intent, suicidal thoughts, and suicidal plans by age 16, with depressive symptoms at age 12 partly mediating this relationship.

Clinical studies reveal even more worrying patterns. For example, in an outpatient sample of autistic youth (n=103; aged 10-17 years), 83.5% reported lifetime suicidal ideation and 24.3% had attempted suicide. Despite this high risk, suicide prevention interventions tailored specifically for autistic individuals are still rare. Importantly, no specialized tools are currently available for autistic youth. To fill this gap, the current study protocol describes the development of a new Visual Safety Plan for Autistic Youth (VSP-AY) and details the plan to assess its effectiveness with autistic adolescents.

The Safety Planning Intervention (SPI) is an evidence-based suicide prevention tool that offers personalized coping strategies, organized into six key steps: (1) recognizing warning signs, (2) using internal coping skills, (3) engaging in social interactions for distraction, (4) contacting supportive individuals, (5) reaching out to mental health providers, and (6) removing lethal means. SPI has proven effective in reducing suicidal behavior and increasing treatment engagement among non-autistic adults. Given this demonstrated effectiveness, SPI has become a core recommended element of clinical practice when suicidal thoughts or behaviors are present and can be incorporated into treatment protocols or used as a standalone intervention.

However, evidence for its effectiveness among adolescents remains limited. A recent meta-analysis of safety planning interventions in adolescents (n = 1,002) found no significant associations with reductions in suicidal ideation, behavior, or attempts. Despite these mixed findings across age groups, SPI's proven effectiveness in adults, combined with the elevated suicide risk among autistic individuals, underscores the importance of examining whether adapted versions could be similarly effective for autistic populations.

Research further shows that developing interventions for autistic individuals needs adaptation because of differences in communication and information processing. Recent efforts have started to address this, with studies pointing out the unique challenges in safety planning with autistic individuals. This has resulted in autism-adapted safety plans for adults and the development of modified assessment tools designed for this group. However, despite this early progress with autistic adults, no evidence-based safety planning interventions have been created or tested specifically for autistic youth.

This gap is particularly concerning, as adolescents display distinctive characteristics regarding suicidal behaviors that differ from adults. Adolescent suicide attempts are often more impulsive, typically involve less lethal methods, and are marked by intentions that are less serious and lethal than those of adults. Additionally, caregiver involvement is crucial in adolescent safety planning, as active parental participation is vital to the process. Yet research indicates that half of autistic youth do not disclose suicidal thoughts to caregivers, while bullying, teasing, and depression emerge as primary precipitants of suicidal behaviors. Together, these findings highlight the need for adaptations that not only address suicide-specific risk factors but also align with the linguistic and visual processing preferences of autistic youth.

Evidence from studies with autistic adults further highlights the need for language adaptations in safety planning. Autistic adults often struggle to identify and express emotions, which requires additional support to effectively engage with safety planning materials. Research also stresses the importance of clear and concrete language to help identify coping strategies. Additionally, terminology changes have been shown to lower distress and improve accessibility, such as reframing "reasons for living" into "what is important to me?" Overall, these findings show that linguistic adaptations are a crucial step in developing effective safety planning interventions for autistic populations.

In addition to these language modifications, research consistently shows that autistic youth respond more effectively to visual stimuli than to verbal communication. Visual channels enable clearer comprehension and more efficient information processing. Visual supports also promote predictability and structure, helping autistic youth create an organized learning environment that reduces anxiety levels. These findings align with recommendations from suicide prevention specialists, who emphasize the importance of visual adaptations in safety planning interventions for autistic youth. Incorporating visual elements into SPI may therefore enhance accessibility, clarity, and engagement, particularly in moments of crisis.

The current research advances the field in two critical ways. First, it focuses specifically on autistic youth aged 13-21 years, a highly vulnerable population that requires tailored interventions. Second, it introduces comprehensive adaptations that integrate both language modifications and visual supports-elements that have not yet been fully combined in existing interventions for this group. The absence of evidence-based SPIs that systematically incorporate both linguistic and visual adaptations represents a key barrier to addressing self-harm and suicidal thoughts and behaviors in autistic youth. This gap underscores the urgent need for developing and evaluating the Visual Safety Plan for Autistic Youth (VSP-AY). The section below describes the co-development process of VSP-AY, which has been completed to enable evaluation of this intervention in the current study.

Intervention Development International Collaboration and Theoretical Framework VSP-AY development resulted from an international partnership involving Israeli researchers and collaborators from the University of Nottingham (UK), La Trobe University, Deakin University (Australia), and Bournemouth University (UK). The development followed the Knowledge-to-Action framework and participatory research principles, with autistic individuals serving as equal partners throughout. The Israeli team formed the Collaborative Research Group for Mental Health and Suicide Prevention among Autistic People, which includes both non-autistic researchers and autistic community experts with lived experience, who act as co-leaders in all research activities. Each project functions through co-leadership pairs-one autistic and one non-autistic researcher-with shared decision-making and joint authorship.

Qualitative Co-development The investigators conducted in-depth interviews with 26 participants: autistic adults with experience of suicide or self-harm (n=16), mental health professionals working with autistic youth (n=10), and parents of autistic youth with a history of suicide or self-harm (n=3). Participants reviewed the UK-developed Autism Adapted Safety Plan (AASP) and provided detailed feedback on clarity, terminology, gaps, and expected responses.

Visual Design Co-development The research team partnered with the Design Department at the College of Management Academic Studies. Design students received comprehensive training on autism characteristics, therapeutic context, suicide prevention principles, and the linguistically adapted protocol. Students participated in iterative design cycles, incorporating feedback from autistic community members, researchers, and supervising designers, resulting in three optimized visual concepts for final selection by an expanded stakeholder group. The development of VSP-AY was based on this multi-stage qualitative process. The current study protocol now focuses on evaluating the finalized Visual Safety Plan for Autistic Youth (VSP-AY) through a pilot randomized controlled trial with two main objectives: (1) to assess its feasibility, usability, and acceptability; and (2) to examine its effectiveness in supporting utilization during crises and in reducing self-injurious and suicidal behaviors among autistic youth.

This study is a pilot randomized controlled trial (RCT) of a visual suicide prevention tool, the Visual Safety Plan for Autistic Youth (VSP-AY). The trial will be conducted in partnership with Geha Mental Health Center, which offers comprehensive mental health services in central Israel and includes both inpatient and outpatient units for adolescents. The center receives many referrals for youth experiencing suicidal thoughts, behaviors, and self-harm, with a significant portion of these involving autistic youth. This makes Geha an ideal setting for recruiting the target population.

Study Design and Methods Setting and Participants The study will recruit 90 autistic youth (45 per group: VSP-AY intervention vs. treatment as usual) through mental health professionals from various disciplines-including psychiatrists, psychologists, social workers, and art therapists-who work directly with autistic youth experiencing suicidal thoughts, behaviors, or self-harm. Eligible participants will be aged 13-18 years (matching the age range served by Geha Mental Health Center's adolescent units), have a formal autism diagnosis, and have experienced suicidal thoughts or behaviors within the past six months. Participants must be able to engage in the study intellectually (either verbally or in writing), not be at imminent risk of suicide, and have adequate family support. Exclusion criteria include immediate suicide risk requiring inpatient care, active psychotic or manic symptoms, and lack of family support as known to social services. Informed consent will be obtained from parents, and assent from adolescents, using documentation designed to be accessible for autistic participants.

Assessments Outcomes are evaluated at three timepoints: baseline (T0) before randomization, post-intervention (T1) when treatment ends (usually 8-12 weeks), and one-month follow-up (T2). Assessments are scheduled prior to regular therapy appointments to reduce burden.

Primary Outcomes - Feasibility Recruitment rate (number recruited divided by approached; target ≥60%), completion rate (percentage completing all procedures; target ≥70%), and dropout rate (percentage withdrawing; target ≤30%). Detailed tracking includes reasons for non-participation, non-completion, and dropout.

Primary Outcomes - Acceptability Satisfaction questionnaires adapted from the Client Satisfaction Questionnaire assess quality, helpfulness, and willingness to recommend, administered to youth, caregivers, and professionals. Semi-structured interviews with purposive samples explore experiences, perceived benefits, challenges, barriers to implementation, and suggestions for improvement. Interviews are analyzed using reflexive thematic analysis conducted collaboratively by autistic and non-autistic researchers.

Secondary Outcomes - Preliminary Effectiveness Columbia Suicide Severity Rating Scale (C-SSRS): Clinician-administered structured interview that assesses suicidal ideation severity (such as wishing to be dead, non-specific thoughts, thoughts with a method, intent without a plan, and intent with a plan), intensity (including frequency, duration, and controllability), and behavior (such as attempts, interrupted or aborted attempts, and preparatory acts) over two weeks.

Non-Suicidal Self-Injury Assessment Tool (NSSI-AT): Evaluates the presence, frequency, methods, and functions of deliberate self-injury without suicidal intent.

Children's Depression Inventory 2nd Edition Self-Report Short Form (CDI 2:SR): a 12-item standardized tool for assessing depressive symptoms in youth aged 7-17, providing scores for Emotional Problems, Functional Problems, and Overall Depression using age/gender-based T-scores.

Ethical Considerations The study will obtain ethical approval from relevant institutional review boards before starting recruitment. Informed consent includes both parental permission and adolescent assent, with accessible procedures for autistic youth (written materials provided in advance, visual aids, concrete language, sufficient processing time). Ongoing consent is stressed, emphasizing the right to withdraw without affecting clinical care. Safety monitoring involves tracking adverse events systematically, referring participants to clinical teams immediately if immediate risk is identified, and conducting monthly safety reviews. Confidentiality is preserved with appropriate limits explained (such as reporting imminent danger, child abuse, or neglect). The participatory approach with autistic co-leaders addresses past concerns about research that is "on" rather than "with" autistic individuals. Dissemination will include accessible formats for diverse audiences and a commitment to develop implementation resources if VSP-AY proves promising.

Significance This research addresses a vital gap by developing and testing the first specialized safety-planning tool for autistic youth. The participatory co-development ensures it is rooted in autistic perspectives while remaining clinically relevant. Results will offer feasibility parameters, acceptability data, and initial effectiveness estimates needed for future large-scale trials, while providing immediate clinical insights for professionals working with suicidal autistic youth. If shown to be feasible, acceptable, and preliminarily effective, VSP-AY could significantly improve suicide prevention services for this vulnerable group worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-18 years
* Formal diagnosis of autism spectrum disorder
* Experienced suicidal ideation or behavior within the past six months
* Able to engage in the study intellectually, either verbally or in writing
* Not at imminent risk of suicide requiring immediate hospitalization
* Have adequate family support
* Able to attend appointments at Geha Mental Health Center
* Parent or legal guardian willing to provide informed consent
* Adolescent willing to provide assent

Exclusion Criteria:

* Immediate suicide risk requiring inpatient hospitalization
* Active psychotic symptoms that prevent meaningful engagement
* Active manic symptoms that prevent meaningful engagement
* Insufficient Hebrew language proficiency to engage with study materials
* Lack of family support, as documented by social services
* Current participation in conflicting intervention studies

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-07-30 (Estimated); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as Measured by Recruitment, Completion, and Dropout Rates | Through study completion, approximately 12 months
  Feasibility is evaluated through three key parameters that assess whether the study can be successfully conducted and whether a future definitive trial is warranted: recruitment rate, completion rate, and dropout rate. Together, these metrics provide essential information about the practicality of conducting a larger-scale efficacy trial.
  Recruitment rate is calculated as the number of participants recruited divided by the number of eligible individuals approached. Detailed tracking includes the number screened, meeting criteria, approached, consenting, and reasons for non-participation. A target of 60% or higher indicates successful recruitment feasibility.
  Completion rate is calculated as the percentage of enrolled participants completing all procedures (baseline, post-intervention, and follow-up assessments). Tracking includes partial completion patterns to identify where attrition occurs. A target of 70% or higher indicates acceptable retention.
  Dropout rate is calculated as the p
Acceptability | Post-intervention (T1, approximately 8-12 weeks) and one-month follow-up (T2)
  Acceptability is evaluated through both quantitative and qualitative methods to comprehensively assess stakeholder perspectives on the Visual Safety Plan for Autistic Youth intervention.
  Satisfaction questionnaires adapted from the Client Satisfaction Questionnaire assess perceived quality, helpfulness, whether the intervention met participant needs, and willingness to recommend the intervention to others or use it again. These questionnaires are administered to youth participants, their caregivers, and mental health professionals who delivered the intervention. Scores range from 8 to 32, with higher scores indicating greater satisfaction.
Acceptability | Post-intervention (T1, approximately 8-12 weeks)
  Semi-structured interviews are conducted with purposive samples of youth participants, caregivers, and professionals to explore experiences in depth. Interview topics include overall experiences with the intervention, perceived benefits and helpful aspects, challenges or difficulties encountered, barriers to implementation, and suggestions for improvement. Interviews are analyzed using a collaborative, reflexive thematic analysis conducted by autistic and non-autistic researchers to identify key themes regarding acceptability and user experience.

SECONDARY OUTCOMES:
Preliminary Effectiveness of Suicidal Ideation | Baseline (T0), Post-intervention (T1, approximately 8-12 weeks), and One-month follow-up (T2)
  Suicidal ideation is assessed using the Columbia Suicide Severity Rating Scale (C-SSRS), a clinician-administered structured interview that evaluates the severity and intensity of suicidal thoughts. The severity subscale assesses the highest level of ideation endorsed over the past two weeks, ranging from passive wish to be dead without specific suicidal thoughts, through increasingly severe levels including non-specific active suicidal thoughts, suicidal thoughts with a method but without intent, suicidal intent without a specific plan, and suicidal intent with a specific plan. Scores range from 0 (no suicidal ideation) to 5 (active suicidal ideation with specific plan and intent), with higher scores indicating more severe ideation. The intensity subscale assesses frequency, duration, controllability, deterrents, and reasons for ideation. The C-SSRS also evaluates suicidal behavior including actual attempts, interrupted attempts, aborted attempts, and preparatory acts.
Preliminary Effectiveness of Non-Suicidal Self-Injury | Baseline (T0), Post-intervention (T1, approximately 8-12 weeks), and One-month follow-up (T2)
  Non-suicidal self-injury is assessed using the Non-Suicidal Self-Injury Assessment Tool (NSSI-AT), which evaluates deliberate self-harm behaviors without suicidal intent. The tool assesses the presence and frequency of NSSI behaviors over the past two weeks, specific methods used such as cutting, scratching, burning, hitting oneself, head-banging, picking at skin or wounds, or interfering with wound healing. The assessment also examines the functions or motivations for NSSI including affect regulation, self-punishment, anti-dissociation, interpersonal influence, anti-suicide, or sensation seeking, as well as contextual factors such as typical locations on the body and situations that precede NSSI episodes. Lower frequency counts indicate improvement in self-injury behaviors.
Preliminary Effectiveness of | Baseline (T0), Post-intervention (T1, approximately 8-12 weeks), and One-month follow-up (T2)
  Depression symptoms are assessed using the Children's Depression Inventory 2nd Edition Self-Report Short Form (CDI 2:SR), a standardized 12-item measure designed for youth aged 7-17 years. The measure evaluates depressive symptoms over the past two weeks across cognitive, affective, and behavioral domains. Each item presents three statements representing increasing severity of a symptom, with participants selecting the statement that best describes their experience. The CDI 2:SR generates three scores: the Emotional Problems subscale, assessing sadness, hopelessness, and anhedonia; the Functional Problems subscale, assessing interpersonal difficulties and school problems; and the Total Depression score, combining all items. Raw scores are converted to T-scores based on age and gender norms, with a mean of 50 and standard deviation of 10. T-scores of 60 or above (84th percentile) indicate elevated symptoms, and T-scores of 70 or above (98th percentile) indicate very elevated symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Geha Mental Health Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the data (mental health information from minors at suicide risk) and ethical obligations to protect participant privacy. This pilot study involves autistic adolescents, a vulnerable population requiring enhanced confidentiality protections. Study results will be disseminated through aggregate findings in peer-reviewed publications, ensuring scientific transparency while maintaining participant confidentiality.

REFERENCES:
- See also: Related Info — https://osf.io/6d59j/overview